CLINICAL TRIAL: NCT00620815
Title: A Phase II, Randomized, Placebo-controlled, Observer-blind, Multi Center Study on the Safety and Immunogenicity of Novartis Tetravalent Influenza Vaccine (Containing Both Interpandemic Strains and H5N1) in Adults Aged 18 Years and Above
Brief Title: Safety and Immunogenicity of Two Doses of a Tetravalent Influenza Vaccine in Adults Aged 18 Years and Above
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V101P1; 2007-002712-25
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Influenza
Keywords: avian flu; seasonal influenza vaccine; influenza vaccine; prepandemic vaccine; virus strain with the potential to cause pandemic; tetravalent vaccine; Prophylaxis of influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- T/P-A (Experimental): One dose of the tetravalent influenza vaccine (T) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by Aflunov (A) on day 22
  Interventions: Biological: MF59-eTIV-H5N1+ placebo /pandemic influenza vaccine
- A/P-T (Experimental): One dose of the Aflunov (A) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by Tetravalent influenza vaccine (T) on day 22.
  Interventions: Biological: Pandemic influenza vaccine + placebo /MF59-eTIV-H5N1
- A/S-A (Active Comparator): One dose of Aflunov (A) and concomitantly, but in a different arm, one dose of licensed seasonal vaccine (S) on day 1, followed Aflunov (A) on day 22.
  Interventions: Biological: Pandemic influenza vaccine + seasonal influenza vaccine /pandemic influenza vaccine
- T/P-A (V2 blood draw) (Experimental): One dose of the tetravalent influenza vaccine (T) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by a blood draw at visit 2 (V2) prior to Aflunov (A) vaccination on day 22.
  Interventions: Biological: MF59-eTIV-H5N1 + Placebo/pandemic influenza vaccine
- A/P-T (V2 blood draw) (Experimental): One dose of the Aflunov(A) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by additional blood draw at visit 2 (V2) prior to the Tetravalent influenza vaccination (T) on day 22.
  Interventions: Biological: Pandemic influenza vaccine + placebo / MF59-eTIV-H5N1
- A/S-A (V2 blood draw) (Active Comparator): One dose of Aflunov (A)and concomitantly, but in a different arm, one dose of licensed seasonal vaccine (S) on day 1, followed by an additional blood draw at visit 2 (V2) prior to Aflunov (A) vaccination on day 22.
  Interventions: Biological: Pandemic influenza vaccine + seasonal influenza vaccine / pandemic influenza vaccine

INTERVENTIONS:
Biological: MF59-eTIV-H5N1+ placebo /pandemic influenza vaccine — Tetravalent influenza vaccine (MF59-eTIV-H5N1)and placebo on day 1 followed 3-5 weeks later by pandemic influenza vaccine, including serology blood draw at V1+V3.
  Arms: T/P-A
Biological: Pandemic influenza vaccine + placebo /MF59-eTIV-H5N1 — Pandemic influenza vaccine plus placebo on day 1 followed 3-5 weeks later by tetravalent influenza vaccine (MF59-eTIV-H5N1), including serology blood draw at V1+V3.
  Arms: A/P-T
Biological: Pandemic influenza vaccine + seasonal influenza vaccine /pandemic influenza vaccine — Pandemic influenza vaccine plus seasonal influenza vaccine, 3-5 weeks later pandemic influenza vaccine , including serology blood draw at V1+V3.
  Arms: A/S-A
Biological: Pandemic influenza vaccine + placebo / MF59-eTIV-H5N1 — Pandemic influenza vaccine plus placebo followed 3-5 weeks later by tetravalent influenza vaccine (MF59-eTIV-H5N1), including serology blood draw at V1, V2 and V3.
  Arms: A/P-T (V2 blood draw)
Biological: Pandemic influenza vaccine + seasonal influenza vaccine / pandemic influenza vaccine — Pandemic influenza vaccine plus seasonal influenza vaccine followed 3-5 weeks later by pandemic influenza vaccine, including serology blood draw at V1, V2 and V3.
  Arms: A/S-A (V2 blood draw)
Biological: MF59-eTIV-H5N1 + Placebo/pandemic influenza vaccine — Tetravalent influenza vaccine (MF59-eTIV-H5N1)plus placebo followed 3-5 weeks later by pandemic influenza vaccine, including serology blood draw at V1, V2 and V3.
  Arms: T/P-A (V2 blood draw)

SUMMARY:
Evaluate the immune response and reactogenicity of H5N1 vaccination in adults aged 18 years and above (as part of a tetravalent vaccine)

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (aged 18 years and above) who have signed an informed consent form

Exclusion Criteria:

* Any acute or chronic illness
* Receipt of seasonal influenza vaccine for the current season 2007/2008
* Known or suspected impairment/alteration of immune function
* Receipt of another vaccine within 3 weeks prior to Visit 1 or planned vaccination within 3 weeks following the last study vaccination
* Any serious disease
* Hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein,neomycin or kanamycin or any other component of the study vaccine
* Receipt of blood, blood products or immunoglobulins 3 months prior to vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis
Locations (2):
- Germany (2):
  - ATRIUM Gesundheitszentrum;, Holzkirchen
  - International Medicine & Public Health Dept. of Infect. Diseases, Munich

REFERENCES:
- [Derived] Herbinger KH, von Sonnenburg F, Nothdurft HD, Perona P, Borkowski A, Fragapane E, Nicolay U, Clemens R. A phase II study of an investigational tetravalent influenza vaccine formulation combining MF59(R): adjuvanted, pre-pandemic, A/H5N1 vaccine and trivalent seasonal influenza vaccine in healthy adults. Hum Vaccin Immunother. 2014;10(1):92-9. doi: 10.4161/hv.26495. Epub 2013 Sep 20. PMID 24047817

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 sites in Germany
Pre-assignment Details: All subjects were included in the trial. The data entered is for the overall study.
Groups:
- T/P-A: one dose of the tetravalent (T) influenza vaccine administered concomitantly, in a different arm, with one dose of the placebo (P) control, on study day 1, followed by Aflunov, on study day 22
- A/P-T: one dose of the Aflunov (A; A/H5N1) avian influenza vaccine administered concomitantly, in a different arm, with one dose of the placebo (P) control, on study day 1, followed by the tetravalent (T) influenza vaccine, on study day 22
- A/S-A: one dose of the Aflunov (A, A/H5N1) avian influenza vaccine administered concomitantly, in a different arm, one dose of licensed seasonal (S) vaccine, on study day 1, followed by Aflunov (A), on study day 22
Period: Overall Study
Arm/Group | T/P-A | A/P-T | A/S-A
Started | 199 | 203 | 199
Completed | 195 | 192 | 192
Not Completed | 4 | 11 | 7
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 6 | 3
Not completed — Inappropriate enrolment | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- A/S-A: one dose of the Aflunov (A; A/H5N1) avian influenza vaccine administered concomitantly, in a different arm, one dose of licensed seasonal(S) vaccine, on study day 1, followed by Aflunov (A), on study day 22
- Total: Total of all reporting groups
Arm/Group | T/P-A | A/P-T | A/S-A | Total
Number analyzed (Participants) | 199 | 203 | 199 | 601
Age, Customized [Number; unit: participants] — A total of 601 subjects were enrolled and randomized, 199 to the T/P-A group, 203 to the A/P-T group and 199 to the A/S-A group. One subject in the A/S-A group did not meet entry criteria and so did not receive any vaccination.
  participants
    ≤60 years | 196 (8) | 202 (9.8) | 198 (9.6) | 596
    ≥ 61 Years | 3 (1) | 1 (0) | 0 (NA) | 4
Sex/Gender, Customized [Number; unit: participants] — Analysis was done on Full Analysis Set
  participants
    Female (≤60 years of age) | 126 | 129 | 114 | 369
    Male (≤60 years of age) | 70 | 73 | 84 | 227
    Female (≥61 years of age) | 1 | 1 | 0 | 2
    Male (≥61 years of age) | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate the Equivalence of Antibody Response Against A/H5N1 Strain Elicited by the Three Different Immunization Schedules on Day 43.
Description: The antibody response was determined by SRH assay. Geometric mean areas (GMAs) and geometric mean ratios (GMRs) in the SRH assay were used to demonstrate the equivalence.
  The statistical analysis was done based on the GMRs.
Time Frame: up to day 43
Population: The analysis was done on Per Protocol Set (PPS)
Measure: Geometric Mean (95% Confidence Interval); unit: Area (mm^2)
Arm/Group | T/P-A | A/P-T | A/S-A
Number analyzed (Participants) | 194 | 202 | 198
Area (mm^2)
  Day 1 | 4.64 [4.17 to 5.17] | 4.10 [3.69 to 4.56] | 4.61 [4.14 to 5.13]
  Day 22 (N= 31, 31, 30) | 14 [10 to 19] | 12 [8.51 to 16] | 16 [12 to 23]
  Day 43 (N=181, 189, 189) | 41 [36 to 47] | 35 [31 to 40] | 39 [34 to 44]
Statistical Analysis 1: Comparison: T/P-A vs A/P-T; (On day 1) Null hypothesis representing non-equivalence was rejected if the two-sided (1-2α)*100% CI on one GMA ratio is completely within the equivalence range [0.5, 2.0]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Group Mean Ratio = 1.13, 96.67% CI 2-sided [1.02 to 1.25]
Statistical Analysis 2: Comparison: T/P-A vs A/S-A; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratios = 1.01, 96.67% CI 2-sided [0.91 to 1.12]
Statistical Analysis 3: Comparison: A/P-T vs A/S-A; (On day 1)Null hypothesis representing non-equivalence was rejected if the two-sided (1-2α)*100% CI on one GMA ratio is completely within the equivalence range [0.5, 2.0]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratio = 0.89, 96.67% CI 2-sided [0.80 to 0.99]
Statistical Analysis 4: Comparison: T/P-A vs A/P-T; (On day 22) Null hypothesis representing non-equivalence was rejected if the two-sided (1-2α)*100% CI on one GMA ratio is completely within the equivalence range [0.5, 2.0]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratios = 1.19, 96.67% CI 2-sided [0.74 to 1.93]
Statistical Analysis 5: Comparison: T/P-A vs A/S-A; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratios = 0.85, 96.67% CI 2-sided [0.52 to 1.38]
Statistical Analysis 6: Comparison: A/P-T vs A/S-A; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratios = 0.71, 96.67% CI 2-sided [0.44 to 1.15]
Statistical Analysis 7: Comparison: T/P-A vs A/P-T; (On day 43) Null hypothesis representing non-equivalence was rejected if the two-sided (1-2α)*100% CI on one GMA ratio is completely within the equivalence range [0.5, 2.0]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratios = 1.14, 96.67% CI 2-sided [1.01 to 1.30]
Statistical Analysis 8: Comparison: T/P-A vs A/S-A; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratios = 1.05, 96.67% CI 2-sided [0.93 to 1.19]
Statistical Analysis 9: Comparison: A/P-T vs A/S-A; [analysis description as in outcome 1, analysis 7]; Test type: Non-Inferiority or Equivalence — To show statistical equivalence was, confidence intervals (CIs) of all 3 pair wise ratios of the GMAs were inspected; ANOVA — P-values were not calculated for the equivalence tests due to lack of appropriate statistical software; Geometric Mean Ratios = 0.92, 96.67% CI 2-sided [0.81 to 1.04]

2. Secondary Outcome: Number of Subjects (Subjects ≤ 60 Years) With Reported Local Reactions After First Vaccination
Description: Local reactions were collected up to 7 days after 1st vaccinations. All subjects were instructed to complete a diary card to record local reactions starting on the day of vaccination (after 6 hours) and for each of the 6 days following each immunization. The table represents local reactions after first vaccination in each arm differently.
Time Frame: Up to 7 days after 1st vaccination
Population: The analysis was performed on Safety Population
Measure: Number; unit: Participants
Groups:
- T/P-A: In Arm Receiving Tetravalent Vaccine (T): Local reactions after first vaccination in arm receiving tetravalent influenza vaccine in group receiving one dose of the tetravalent influenza vaccine (T) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by Aflunov (A) on day 22
- T/P-A: In Arm Receiving Placebo (P): Local reactions after first vaccination in arm receiving placebo in group receiving one dose of the tetravalent influenza vaccine (T) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by Aflunov (A) on day 22
- A/P-T: In Arm Receiving Aflunov (A): Local reactions after first vaccination in arm receiving Aflunov in group receiving one dose of the Aflunov (A) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by Tetravalent influenza vaccine(T) on day 22
- A/P-T: In Arm Receiving Placebo (P): Local reactions after first vaccination in arm receiving Placebo in group receiving one dose of the Aflunov (A) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed by Tetravalent influenza vaccine (T) on day 22
- A/S-A: In Arm Receiving Aflunov (A): Local reactions after first vaccination in arm receiving Aflunov in group receiving one dose of Aflunov (A) and concomitantly, but in a different arm, one dose of licensed seasonal vaccine (S) on day 1, followed Aflunov (A) bon day 22
- A/S-A: In Arm Receiving Seasonal Influenza Vaccine (S): Local reactions after first vaccination in arm receiving seasonal influenza vaccination in group receiving one dose of Aflunov (A) and concomitantly, but in a different arm, one dose of licensed seasonal vaccine (S) on day 1, followed Aflunov (A) on day 22
Arm/Group | T/P-A: In Arm Receiving Tetravalent Vaccine (T) | T/P-A: In Arm Receiving Placebo (P) | A/P-T: In Arm Receiving Aflunov (A) | A/P-T: In Arm Receiving Placebo (P) | A/S-A: In Arm Receiving Aflunov (A) | A/S-A: In Arm Receiving Seasonal Influenza Vaccine (S)
Number analyzed (Participants) | 195 | 194 | 201 | 201 | 197 | 196
Participants
  Erythema | 10 | 0 | 5 | 0 | 6 | 5
  Induration | 22 | 1 | 5 | 0 | 9 | 3
  Swelling | 19 | 1 | 6 | 0 | 7 | 3
  Ecchymosis | 2 | 1 | 2 | 0 | 2 | 1
  Pain | 164 | 30 | 138 | 32 | 131 | 80

3. Secondary Outcome: Number of Subjects (Subjects ≤60 Years) With Reported Local Reactions After Second Vaccination
Description: Local reactions were collected up to 7 days after 1st vaccinations. All subjects were instructed to complete a diary card to record local reactions starting on the day of vaccination (after 6 hours) and for each of the 6 days following each immunization.
Time Frame: Up to 7 days after 2nd vaccination
Population: The analysis was performed on Safety Population
Measure: Number; unit: Participants
Groups:
- A/S-A: one dose of the Aflunov (A, A/H5N1) avian influenza vaccine administered concomitantly, in a different arm, one dose of licensed seasonal(S) vaccine, on study day 1, followed by Aflunov (A), on study day 22
Arm/Group | T/P-A | A/P-T | A/S-A
Number analyzed (Participants) | 188 | 192 | 192
Participants
  Erythema (N=188,192,191) | 2 | 7 | 5
  Induration | 7 | 10 | 7
  Swelling | 5 | 8 | 6
  Ecchymosis | 3 | 3 | 2
  Pain | 98 | 136 | 91

4. Secondary Outcome: Number of Subjects (Subjects ≤ 60 Years) With Reported Systemic Reactions After 1st and 2nd Vaccinations.
Description: Systemic reactions were collected upto 7 days after 1st and 2nd vaccinations. All subjects were instructed to complete a diary card to record systemic reactions starting on the day of vaccination (after 6 hours) and for each of the 6 days following each immunization.
Time Frame: 7 days after 1st and 2nd vaccinations each
Population: The analysis was performed on Per Protocol Safety Population
Measure: Number; unit: Participants
Groups:
- T/P-A: After 1st Vaccination: Systemic reactions after first vaccination after one dose of the tetravalent influenza vaccine (T) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed 3 to 5 weeks later by Aflunov (A)
- A/P-T: After 1st Vaccination: Systemic reactions after first vaccination after one dose of Aflunov (A) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed 3 to 5 weeks later by tetravalent influenza vaccine (T)
- A/S-A: After 1st Vaccination: Systemic reactions after first vaccination after one dose of Aflunov (A) and concomitantly, but in a different arm, one dose of licensed seasonal vaccine (S) on day 1, followed 3 to 5 weeks later by Aflunov (A)
- T/P-A: After 2nd Vaccination: Systemic reactions after second vaccination after one dose of the tetravalent influenza vaccine (T) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed 3 to 5 weeks later by Aflunov (A)
- A/P-T: After 2nd Vaccination: Systemic reactions after second vaccination after one dose of Aflunov (A) and concomitantly, but in a different arm, one dose of placebo (P) on day 1, followed 3 to 5 weeks later by tetravalent influenza vaccine (T)
- A/S-A: After 2nd Vaccination: Systemic reactions after second vaccination after one dose of Aflunov (A) and concomitantly, but in a different arm, one dose of licensed seasonal vaccine (S) on day 1, followed 3 to 5 weeks later by Aflunov (A)
Arm/Group | T/P-A: After 1st Vaccination | A/P-T: After 1st Vaccination | A/S-A: After 1st Vaccination | T/P-A: After 2nd Vaccination | A/P-T: After 2nd Vaccination | A/S-A: After 2nd Vaccination
Number analyzed (Participants) | 195 | 201 | 196 | 188 | 192 | 192
Participants
  Chills (N=195,201,196,187,192,192) | 24 | 8 | 9 | 6 | 11 | 3
  Malaise (N=195,201,196,187,192,192) | 62 | 29 | 28 | 15 | 38 | 15
  Myalgia (N=195,201,196,187,192,192) | 68 | 47 | 42 | 22 | 53 | 27
  Arthralgia (N=195,201,196,187,192,192) | 34 | 14 | 12 | 6 | 15 | 6
  Headache (N=195, 201, 196, 187, 192, 192) | 70 | 52 | 43 | 33 | 50 | 27
  Sweating (N=195,201,196,187,192,192) | 13 | 16 | 10 | 6 | 13 | 7
  Fatigue (N=195,201,196,187,192,192) | 79 | 58 | 52 | 32 | 60 | 35
  Nausea (N=195,201,196,187,192,192) | 24 | 16 | 8 | 7 | 16 | 6
  Coughing (N=195,201,196,187,192,192) | 14 | 16 | 16 | 13 | 12 | 13
  Fever (>= 38 C) [N=195,201,195,188,192,192] | 8 | 1 | 3 | 2 | 5 | 0
  Body Temp. (< 38C)[N=195,201,195,188,192,192] | 187 | 200 | 192 | 186 | 187 | 192
  Stayed home due to reactions | 8 | 7 | 2 | 1 | 8 | 1
  Analgesic, Antipyretic Medicines Used | 27 | 21 | 15 | 6 | 16 | 6

5. Secondary Outcome: Percentages of Subjects Achieving Seroconversion/Significant Increase in Antibody Titre/ Area as Measured by SRH and (HI) and at Least 4 Fold Rise in Titres by Micro-neutralization (MN) Assay-H5N1 Strain
Description: Measurement of immunogenicity in terms of significant increase in antibody titer and Seroconversion.
  Significant increase in antibody titer is defined as at least a four-fold increase from non-negative pre-vaccination serum (≥ 10) for HI or a 50% increase in area for SRH.
  Seroconversion is defined as negative pre-vaccination serum / post-vaccination titer ≥40 for HI (area ≥25 mm2 for SRH)
Time Frame: up to day 43
Population: The population was analyzed on per protocol set.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | T/P-A | A/P-T | A/S-A
Number analyzed (Participants) | 181 | 189 | 189
Percentage of subjects
  Seroconversion/significant rise SRH(N=181,189,189) | 90 [84 to 94] | 86 [80 to 90] | 86 [80 to 91]
  Seroconversion/significant rise HI (N=180,186,184) | 69 [62 to 76] | 67 [59 to 73] | 75 [68 to 81]
  Four fold increase MN (N=181,189,189) | 90 [84 to 94] | 86 [80 to 90] | 89 [84 to 93]

6. Secondary Outcome: Percentages of Subjects Achieving HI/MN ≥ 1:40 and SRH Area ≥ 25^mm2
Description: Measurement of immunogenicity in terms of percentage of subjects achieving a titre ≥ 40/area ≥ 25mm^2 after immunization as determined by HI (Haemagglutination Inhibition), MN(Microneutralization) and SRH assay.
Time Frame: Up to 43 days
Population: The analysis was done on Per Protocol Set
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | T/P-A | A/P-T | A/S-A
Number analyzed (Participants) | 196 | 202 | 198
Percentages of subjects
  SRH-Day 1 (N=194,202,198) | 4 [1 to 7] | 0 [0 to 2] | 4 [2 to 8]
  SRH-Day 43 (N=181,189,189) | 93 [88 to 96] | 86 [80 to 90] | 89 [84 to 93]
  HI-Day 1 (N=192,198,193) | 2 [0 to 4] | 0 [0 to 2] | 2 [0 to 4]
  HI-Day 43 (N=181,187,186) | 70 [62 to 76] | 66 [59 to 73] | 74 [67 to 80]
  MN-Day 1 (N=194,202,198) | 1 [0 to 4] | 3 [1 to 6] | 3 [1 to 6]
  MN-Day 43 (N=181,189,189) | 90 [85 to 94] | 87 [82 to 92] | 89 [84 to 93]

7. Secondary Outcome: Antibody Response Determined by HI and MN Assay.
Description: Measurement of immunogenicity in terms of Geometric mean titers (GMTs) as determined by HI and MN assay.
Time Frame: Up to 43 days
Population: The population was analyzed on Per protocol set
Measure: Mean (95% Confidence Interval); unit: titers
Arm/Group | T/P-A | A/P-T | A/S-A
Number analyzed (Participants) | 192 | 198 | 193
titers
  HI-Day 1 | 5.93 [5.49 to 6.40] | 5.58 [5.18 to 6.02] | 5.85 [5.42 to 6.32]
  HI-Day 22 (N=31,31,30) | 8.36 [5.79 to 12] | 6.76 [4.68 to 9.77] | 9.66 [6.65 to 14]
  HI-Day 43 (N=181,187,186) | 46 [30 to 70] | 33 [22 to 50] | 49 [32 to 75]
  MN-Day 1 (N=194,202,198) | 10 [9.28 to 11] | 10 [9.67 to 11] | 10 [9.55 to 11]
  MN-Day 22 (N=31,31,30) | 14 [11 to 19] | 16 [12 to 22] | 17 [13 to 23]
  MN-Day 43 (N=181,189,189) | 141 [110 to 180] | 111 [87 to 141] | 133 [105 to 169]

8. Secondary Outcome: Percentages of B-cell Antibodies Against H5N1 and H1N1 After Each Vaccination.
Description: The Cell Mediated Immunity (CMI) response was evaluated in a randomly selected subgroup of approximately 92 subjects from all the vaccine groups out of a total of 601 enrolled subjects.
  Frequency of circulating memory B cells (MBC), capable of differentiating in vitro into cell secreting IgG (Immunoglobulin G) antibodies specific for H5N1 (the subunit from A/Vietnam/1194/2004) or for H1N1 (the subunit from A/Solomon Island/3/2006) were determined by an ELISA-coupled limiting dilution assay.The frequency of H5N1-IgG MBC and H1N1-IgG MBC was expressed as percentages (%) of total IgG producing MBC.
Time Frame: Three weeks after first vaccination (day 22) and three weeks after second vaccination (day 43)
Population: The analysis was done on Full analysis set
Measure: Mean (95% Confidence Interval); unit: Percentages of B-cell antibodies
Arm/Group | T/P-A | A/P-T | A/S-A
Number analyzed (Participants) | 30 | 30 | 29
Percentages of B-cell antibodies
  H5N1-IgG MBC - Day 1 (N=30, 30, 29) | 0.7 [0.11 to 1.28] | 0.42 [-0.168 to 1.01] | 0.53 [-0.073 to 1.12]
  H5N1-IgG MBC - Day 22 (N=30, 30, 28) | 5.39 [2.66 to 8.11] | 6.08 [3.36 to 8.8] | 7.58 [4.77 to 10]
  H5N1-IgG MBC - Day 43 (N=30, 30, 29) | 6.67 [4.71 to 8.64] | 7.21 [5.24 to 9.18] | 6.84 [4.84 to 8.83]
  H1N1-IgG MBC - Day 1 (N=30, 30, 29) | 2.35 [0.81 to 3.89] | 2.64 [1.1 to 4.18] | 1.61 [0.039 to 3.18]
  H1N1-IgG MBC - Day 22 (N=30, 30, 28) | 13 [9.29 to 17] | 8.55 [4.76 to 12] | 15 [11 to 19]
  H1N1-IgG MBC - Day 43 (N=30, 30, 29) | 12 [6.98 to 17] | 16 [11 to 21] | 15 [10 to 20]

9. Secondary Outcome: Mean T-Cells Per Million Total Cells (95% CI) in Response to H5 Peptides and H5N1 Subunit
Description: Frequency and functionality of vaccine antigen-specific CD4+ (cluster of differentiation 4) T cells was assessed in peripheral blood (PBMC) taken at days 1, 22 and 43 after in vitro stimulation with:
  Library of 70 peptides spanning the whole H5 A/Vietnam/1194/2004 protein (H5 pool of 70 Vietnam) H5N1 subunit from A/Vietnam/1194/2004 (H5N1 Vietnam) H3N2 subunit from A/ Wisconsin/67/2005 (H3N2 Wisconsin) H1N1 subunit from A/Solomon Islands/3/2006 (H1N1 Solomon Islands) Polyclonal stimulus agonistic aCD3 mAb [monoclonal antibody (aCD3)].
  The change in frequency of T-cells was measured.
Time Frame: Three weeks after 1st vaccination (day 22) and three weeks after 2nd vaccination (day 43)
Population: Analysis was done on full analysis set
Measure: Mean (95% Confidence Interval); unit: Mean cells per million total cells
Arm/Group | T/P-A | A/P-T | A/S-A
Number analyzed (Participants) | 31 | 31 | 30
Mean cells per million total cells
  H5 Pool of 70 Vietnam Day 1 (N=30, 31, 30) | 162 [106 to 218] | 175 [120 to 230] | 167 [111 to 223]
  H5 Pool of 70 Vietnam Day 22 (N=31, 31, 30) | 273 [198 to 348] | 358 [284 to 431] | 365 [290 to 440]
  H5 Pool of 70 Vietnam Day 43 (N=31, 31, 30) | 311 [246 to 376] | 328 [264 to 392] | 290 [225 to 355]
  H5N1 Vietnam Day 1 (N=31, 31, 30) | 136 [93 to 178] | 180 [137 to 222] | 155 [112 to 198]
  H5N1 Vietnam Day 22 (N=31, 31, 30) | 604 [420 to 788] | 711 [526 to 895] | 938 [752 to 1124]
  H5N1 Vietnam Day 43 (N=31, 31, 30) | 784 [615 to 952] | 813 [644 to 982] | 750 [579 to 921]
  H3N2 Wisconsin Day 1 (N=31, 31, 30) | 329 [266 to 392] | 344 [281 to 407] | 349 [285 to 413]
  H3N2 Wisconsin Day 22 (N=31, 31, 30) | 1050 [853 to 1247] | 616 [419 to 813] | 1129 [929 to 1329]
  H3N2 Wisconsin Day 43 (N=31, 31, 30) | 910 [750 to 1071] | 1034 [874 to 1195] | 814 [651 to 978]
  H1N1 Solomon Islands Day 1 (N=30, 31, 30) | 275 [186 to 365] | 427 [339 to 515] | 331 [241 to 420]
  H1N1 Solomon Islands Day 22 (N=30, 30, 30) | 998 [795 to 1201] | 729 [528 to 930] | 1040 [842 to 1237]
  H1N1 Solomon Islands Day 43 (N=30, 30, 29) | 930 [735 to 1125] | 973 [781 to 1166] | 792 [599 to 984]
  aCD3 Day 1 (N=31, 31, 30) | 38714 [29922 to 47505] | 32703 [23912 to 41494] | 27824 [18887 to 36760]
  aCD3 Day 22 (N=31, 31, 30) | 29134 [26356 to 31911] | 27324 [24571 to 30077] | 32324 [29504 to 35144]
  aCD3 Day 43 (N=31, 31, 30) | 31001 [27850 to 34153] | 29327 [26203 to 32451] | 34680 [31480 to 37880]

ADVERSE EVENTS:
Time Frame: Throughout the entire study period
Description: Data provided in the "other Adverse Events (>5%)" includes solicited local and systemic reactions along with unsolicited Adverse Events (AEs) that persisted for more than 7 days after each study vaccination. Events not otherwise noted as occurring in the >= 61 year old population were limited to the <= 60 year old population.
Arm/Group | T/P-A | A/P-T | A/S-A
Serious Adverse Events (participants affected / at risk) | 2/199 | 3/203 | 4/198
Other Adverse Events (participants affected / at risk) | 190/199 | 185/203 | 183/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T/P-A (N=199) | A/P-T (N=203) | A/S-A (N=198)
Retinal Detachment (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Polyp (Gastrointestinal disorders) | 1 | 0 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Endoscopic Retrograde Cholangiopancreatography (Investigations) | 0 | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 0 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Bulimia Nervosa (Psychiatric disorders) | 0 | 0 | 1
Depression Suicidal (Psychiatric disorders) | 0 | 0 | 1
Eye Operation (Surgical and medical procedures) | 0 | 1 | 0
Hysterosalpingo-Oophorectomy (Surgical and medical procedures) | 0 | 0 | 1
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | T/P-A (N=199) | A/P-T (N=203) | A/S-A (N=198)
Nausea (Gastrointestinal disorders) | 30 | 29 | 14
Chills (General disorders) | 30 | 19 | 11
Injection Site Erythema (General disorders) | 10 | 10 | 11
Injection Site Haemorrhage (General disorders) | 13 | 11 | 8
Injection Site Induration (General disorders) | 22 | 14 | 12
Injection Site Pain (General disorders) | 172 | 164 | 155
Injection Site Swelling (General disorders) | 21 | 12 | 11
Malaise (General disorders) | 66 | 55 | 38
Pyrexia (General disorders) | 12 | 11 | 6
Nasopharyngitis (Infections and infestations) | 39 | 38 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 29 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 75 | 77 | 57
Headache (Nervous system disorders) | 90 | 86 | 60
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 28 | 26
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 19 | 25 | 15
Diarrhoea (Gastrointestinal disorders) | 9 | 11 | 9
Toothache (Gastrointestinal disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Fatigue (General disorders) | 1/3 | 1/1 | 0/0 — In subjects >= 61 years of age.
Injection Site Haematoma (General disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Injection Site Haemorrhage (General disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Injection Site Pain (General disorders) | 2/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Malaise (General disorders) | 1/3 | 1/1 | 0/0 — In subjects >= 61 years of age.
Nasopharyngitis (Infections and infestations) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Tinea Pedis (Infections and infestations) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/3 | 1/1 | 0/0 — In subjects >= 61 years of age.
Back Pain (Musculoskeletal and connective tissue disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Myalgia (Musculoskeletal and connective tissue disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Headache (Nervous system disorders) | 1/3 | 1/1 | 0/0 — In subjects >= 61 years of age.
Cough (Respiratory, thoracic and mediastinal disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Wisdom teeth Removal (Surgical and medical procedures) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/3 | 0/1 | 0/0 — In subjects >= 61 years of age.
Fatigue (General disorders) | 88 | 92 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days